CLINICAL TRIAL: NCT05468736
Title: A Phase 2/3 Age De-escalating Study to Evaluate the Safety and Immunogenicity of a SARS-CoV-2 Recombinant Spike Protein Vaccine (SARS-CoV-2 rS) With Matrix-M™ Adjuvant in Children 6 Months to < 12 Years of Age
Brief Title: Study to Evaluate Safety and Immunogenicity of COVID-19 Vaccine in Children 6 Months to < 12 Years
Acronym: COVID-19
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019nCoV-503
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — NVX-CoV2373 adjuvated lipid nanoparticle; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Cohort-1(6 to < 12 y)-Part-1(Active Vaccine) (Experimental): NVX-CoV2373 (SARS-CoV-2 rS: 5 µg + Matrix-M adjuvant: 50 µg in 0.5 mL)
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Initial Vaccination Period)
- Cohort-1(6 to < 12 y)-Part-1(Placebo) (Placebo Comparator): Placebo (normal saline)
  Interventions: Other: Placebo
- Cohort-1(6 to < 12 y)-Part-2(Active Vaccine) (Experimental): NVX-CoV2373 (SARS-CoV-2 rS: 5 µg + Matrix-M adjuvant: 50 µg in 0.5 mL)
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Initial Vaccination Period)
- Cohort-1(6 to < 12 y)-Part-2(Placebo) (Placebo Comparator): Placebo (normal saline)
  Interventions: Other: Placebo
- Cohort-2(2 to < 6 y)-Part-1(Active Vaccine) (Experimental): NVX-CoV2373 (SARS-CoV-2 rS: 5 µg + Matrix-M adjuvant: 50 µg in 0.5 mL)
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Initial Vaccination Period)
- Cohort-2(2 to < 6 y)-Part-1(Placebo) (Placebo Comparator): Placebo (normal saline)
  Interventions: Other: Placebo
- Cohort-2(2 to < 6 y)-Part-2(Active Vaccine) (Experimental): NVX-CoV2373 (SARS-CoV-2 rS: 5 µg + Matrix-M adjuvant: 50 µg in 0.5 mL)
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Initial Vaccination Period)
- Cohort-2(2 to < 6 y)-Part-2(Placebo) (Placebo Comparator): Placebo (normal saline)
  Interventions: Other: Placebo
- Cohort-3(6 to < 24 m)-Part-1(Active Vaccine) (Experimental): NVX-CoV2373 (SARS-CoV-2 rS: 5 µg + Matrix-M adjuvant: 50 µg in 0.5 mL)
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Initial Vaccination Period)
- Cohort-3(6 to < 24 m)-Part-1(Placebo) (Placebo Comparator): Placebo (normal saline)
  Interventions: Other: Placebo
- Cohort-3(6 to < 24 m)-Part-2 (Experimental): NVX-CoV2373 (SARS-CoV-2 rS: 5 µg + Matrix-M adjuvant: 50 µg in 0.5 mL)
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Initial Vaccination Period)
- Cohort-3(6 to < 24 m)-Part-2(Placebo) (Placebo Comparator): Placebo (normal saline)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Initial Vaccination Period) — Alternating intramuscular (deltoid) injections of SARS-CoV-2 rS co-formulated with Matrix-M1 adjuvant (0.5 mL) (or fractional dose if necessary) on Days 0 and 21 in the Initial Vaccination Period.
  Other Names: NVX-CoV2373
  Arms: Cohort-1(6 to < 12 y)-Part-1(Active Vaccine); Cohort-1(6 to < 12 y)-Part-2(Active Vaccine); Cohort-2(2 to < 6 y)-Part-1(Active Vaccine); Cohort-2(2 to < 6 y)-Part-2(Active Vaccine); Cohort-3(6 to < 24 m)-Part-1(Active Vaccine); Cohort-3(6 to < 24 m)-Part-2
Other: Placebo — Alternating intramuscular (deltoid) injections of placebo (0.5 mL) on Days 0 and 21 in the Initial Vaccination Period or on Days 201 or Day 229 in the Booster Vaccination Period
  Other Names: Sodium chloride 0.9% (BP, sterile)
  Arms: Cohort-1(6 to < 12 y)-Part-1(Placebo); Cohort-1(6 to < 12 y)-Part-2(Placebo); Cohort-2(2 to < 6 y)-Part-1(Placebo); Cohort-2(2 to < 6 y)-Part-2(Placebo); Cohort-3(6 to < 24 m)-Part-1(Placebo); Cohort-3(6 to < 24 m)-Part-2(Placebo)

SUMMARY:
This is a Phase 2/3 randomized, observer-blinded, placebo-controlled, age de-escalation trial to evaluate the safety and immunogenicity of 2 primary doses of SARS-CoV-2 rS with Matrix-M™ adjuvant (NVX-CoV2373) given 21 days apart and NVX CoV2373 or a variant-based vaccine given as a booster dose or at crossover in pediatric participants (3 age cohorts; 6 to < 12 years, 2 to < 6 years, and 6 to < 24 months of age). Each age cohort will be conducted in 2 parts starting with the oldest age cohort (6 to < 12 years of age).

DETAILED DESCRIPTION:
This is a Phase 2/3 randomized, observer-blinded, placebo-controlled, age de-escalation trial to evaluate the safety and immunogenicity of 2 primary doses of SARS-CoV-2 rS with Matrix-M™ adjuvant (NVX-CoV2373) given 21 days apart and NVX CoV2373 or a variant-based vaccine given as a booster dose or at crossover in pediatric participants (3 age cohorts; 6 to < 12 years, 2 to < 6 years, and 6 to < 24 months of age).

Each age cohort will be conducted in 2 parts starting with the oldest age cohort (6 to < 12 years of age).

Part 1 will enroll approximately 120 healthy or medically stable sentinel participants per age cohort (10% of the intended enrollment population per age cohort, for a total of 360 sentinel participants overall) who will be randomized in a 1:1 ratio to receive 2 doses of NVX-CoV2373 or placebo with doses given 21 days apart.

Part 2 will enroll a larger number of healthy or medically stable participants (N= approximately 1,080 per age cohort), for a total of approximately 3,240 pediatric participants enrolled in Part 2, and a total of approximately 3,600 participants enrolled in the entire trial). Initial randomization in Part 2 will be in a 2:1 ratio, and the safety and effectiveness of 2 doses of NVX-CoV2373 given 21 days apart will be assessed.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, each individual must satisfy all of the following criteria:

1. Pediatric participants 6 months to < 12 years of age at randomization, determined to be healthy or medically stable by the investigator (based on review of health status, vital signs [to include body temperature], medical history, and targeted physical examination [to include body weight]). Vital signs must be within the normal range prior to the first vaccination, according to the child's age, sex, weight, and height/length.
2. For children from 6 months to < 12 months of age: born at full-term (≥ 37 weeks gestation) with a minimum birth weight of 2.5 kilograms (kg).
3. Participant and parent(s)/caregiver(s) or legally acceptable representative willing and able to give informed consent and assent, as required, prior to study enrollment and to comply with study procedures.
4. Participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through 3 months after the last vaccination OR agree to consistently use a highly effective contraception method from at least 28 days prior to enrollment and through 3 months after the last vaccination.
5. Agree not to participate in another SARS-CoV-2 prevention trial for the duration of the study.

Exclusion Criteria:

If an individual meets any of the following criteria, he or she is ineligible for this study:

1. Any acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4°F [≥ 38.0°C]). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided.
2. Unstable acute or chronic illness. Criteria for unstable medical conditions include:

   1. Substantive changes in chronic prescribed medication (change in class or significant change in dose) in the past 2 months.
   2. Currently undergoing workup of undiagnosed illness that could lead to a diagnosis of a new condition.

   NOTE: Well-controlled human immunodeficiency virus [HIV] infection with undetectable HIV ribonucleic acid [RNA < 50 copies/mL] and CD4 count > 200 cells/µL for at least 1 year, documented within the last 6 months, is NOT considered an unstable chronic illness. Participant's or parent's/caregiver's verbal report will suffice as documentation.
3. Participation in research involving an investigational product (drug/biologic/device) administered within 45 days prior to the first study vaccination.
4. History of a previous laboratory-confirmed diagnosis of SARS-CoV-2 infection or COVID-19.
5. Prior administration of an investigational, authorized, or approved Coronavirus vaccine (ie, against either SARS-CoV, SARS-CoV-2, or MERS CoV) or expected receipt during the period of study follow-up.
6. Previous or current diagnosis of MIS-C.
7. Receipt of medications intended to prevent or treat COVID-19.
8. Received any vaccine within 14 days prior to first study vaccination or planned receipt of any vaccine before Day 49 (ie, 28 days after the second vaccination), except for influenza vaccination, which may be received > 14 days prior to or > 14 days after any study vaccination.
9. Known or suspected congenital or acquired immunodeficiency or autoimmune disease/condition; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (prednisone or equivalent for > 14 continuous days) within 90 days prior to first study vaccination. NOTE: An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 20 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids is permitted. Topical tacrolimus and ocular cyclosporin are permitted. Stable autoimmune endocrine disorders (eg, thyroiditis, pancreatitis), including stable diabetes mellitus type 1, or participants with a history of Kawasaki disease are NOT excluded.
10. Received immunoglobulin or blood-derived products within 90 days prior to first study vaccination.
11. Active cancer (malignancy) on chemotherapy within 1 year prior to first study vaccination (with the exception of malignancy cured via excision, at the discretion of the investigator).
12. Any known allergies to products contained in the investigational product.
13. Participants who are breastfeeding a child, pregnant or who plan to become pregnant within 3 months following the last study vaccination.
14. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with the evaluation of the trial vaccine or interpretation of study results.
15. Study team member or first-degree relative of any study team member (inclusive of Sponsor, and study site personnel involved in the study).
16. Current participation in any other COVID-19 prevention clinical trial.
17. Participants with a history of myocarditis or pericarditis.

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3600 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Reactogenicity Incidence and Severity | Day 0 to Day 7
  Reactogenicity incidence, duration, and severity (mild, moderate, severe, or potentially life-threatening) recorded by parent(s)/caregiver(s) on an electronic patient-reported outcome diary application (eDiary) on days of vaccination and subsequent 6 days (total 7 days after each vaccine injection).
Incidence and Severity of Medically Attended Adverse Events (MAAEs) | Day 0 to Day 28
  Incidence and severity of MAAEs through 28 days after second injection of each set of vaccinations (initial and crossover), and after a booster dose.
Incidence and Severity of Unsolicited Adverse Events (AEs) | Day 0 to Day 28
  Incidence and severity of unsolicited AEs through 28 days after second injection of each set of vaccinations (initial and crossover), and after a booster dose.
Incidence and Severity of MAAEs Attributed to Study Vaccine | Day 0 to Day 730
  Incidence and severity of MAAEs attributed to study vaccine after initial vaccination at Day 0 through Month 24 or the EoS.
Incidence and Severity of Serious Adverse Events (SAEs) | Day 0 to Day 730
  Incidence and severity of SAEs after initial vaccination at Day 0 through Month 24 or the EoS.
Incidence and Severity of Adverse Events of Special Interest (AESIs) | Day 0 to Day 730
  Incidence and severity of AESIs (including multisystem inflammatory syndrome in children [MIS-C], and myocarditis and/or pericarditis) after initial vaccination at Day 0 through Month 24 or the EoS.
Death due to any cause | Day 0 to Day 730
  Death due to any cause occurring from Day 0 to EoS.

SECONDARY OUTCOMES:
Participants with PCR positive mild, moderate or severe COVID-19 after the primary series of 2 doses | Day 0 to Day 730
  Incidence rate of participants with first episode of PCR-positive mild, moderate, or severe COVID-19 overall and per age cohort, with or without positive anti-NP serology at baseline after the primary series of 2 doses.
Participants with PCR positive moderate or severe COVID-19 after the primary series of 2 doses | Day 0 to Day 730
  Incidence rate of participants with first episode of PCR-positive moderate or severe COVID-19 overall and per age cohort, with or without positive anti-NP serology at baseline, and by risk factors to develop severe COVID-19 after the primary series of 2 doses.
Participants with diagnostic test - positive asymptomatic, mild, moderate or severe COVID-19 after the primary series of 2 doses | Day 0 to Day 730
  Incidence rate of participants with first episode of diagnostic test-positive asymptomatic, mild, moderate, or severe COVID-19 (regardless of confirmatory test used, ie, PCR or rapid antigen test, and of testing location, ie, central or externally tested) overall and per age cohort, with or without positive anti-NP serology at baseline after the primary series of 2 doses.
Participants with diagnostic test - positive moderate or severe COVID-19 after the primary series of 2 doses | Day 0 to Day 730
  Incidence rate of participants with first episode of diagnostic test-positive moderate or severe COVID-19 (regardless of confirmatory test used, ie, PCR or rapid antigen test, and of testing location, ie, central or externally tested) overall and per age cohort, with or without positive anti NP serology at baseline, and by risk factors to develop severe COVID-19 after the primary series of 2 doses.
Participants with PCR positive mild, moderate or severe COVID-19 after the booster dose | Day 0 to Day 730
  Incidence rate of participants with first episode of PCR-positive mild, moderate, or severe COVID-19 overall and per age cohort, with or without positive anti-NP serology at baseline after the booster dose.
Participants with PCR positive moderate or severe COVID-19 after the booster dose | Day 0 to Day 730
  Incidence rate of participants with first episode of PCR-positive moderate or severe COVID-19 overall and per age cohort, with or without positive anti-NP serology at baseline, and by risk factors to develop severe COVID-19 after the booster dose.
Participants with diagnostic test - positive asymptomatic, mild, moderate or severe COVID-19 after the booster dose | Day 0 to Day 730
  Incidence rate of participants with first episode of diagnostic test-positive asymptomatic, mild, moderate, or severe COVID-19 (regardless of confirmatory test used, ie, PCR or rapid antigen test, and of testing location, ie, central or externally tested) overall and per age cohort, with or without positive anti-NP serology at baseline after the booster dose.
Participants with diagnostic test moderate or severe COVID-19 after the booster dose | Day 0 to Day 730
  Incidence rate of participants with first episode of diagnostic test-positive moderate or severe COVID-19 (regardless of confirmatory test used, ie, PCR or rapid antigen test, and of testing location, ie, central or externally tested) overall and per age cohort, with or without positive anti-NP serology at baseline after the booster dose, and by risk factors to develop severe COVID-19.
Antibodies to SARS-CoV-2 Nucleoprotein (NP) at Specified Time Points | Day 0 to Day 730
  Antibodies to SARS-CoV-2 NP, regardless of whether the infection was symptomatic. Antibodies to SARS-CoV-2 NP at Days 0 and 35, at Crossover Visit 1, at Booster vaccination visit, and at Months 12 and 24 will be used to determine natural infection and to determine the incidence of asymptomatic infection acquired during study follow-up.
Neutralizing antibody response, post-booster, by age cohort,seronegative to anti-SARS-CoV-2 NP antibodies at baseline and pre-booster | Day 0 to Day 28
  Neutralizing antibody response at 28 days post booster for pediatric participants in the Immunogenicity Population overall and by age cohort, seronegative to anti-SARS-CoV-2 NP antibodies at baseline and pre-booster, compared with that observed at 28 days post-booster vaccination in young adult participants 18 to < 26 years of age.
Neutralizing antibody response, by age cohort, regardless of serostatus at baseline and pre-booster | Day 0 to Day 28
  Neutralizing antibody response at 28 days post-booster for pediatric participants in the Immunogenicity Population overall and by age cohort, regardless of serostatus at baseline and pre-booster, compared with that observed in pediatric participants at baseline (Day 0).
Serum IgG levels to SARS-CoV-2 S protein, post-booster, by age cohort, regardless of serostatus at baseline and pre-booster vaccination | Day 0 to Day 28
  Serum IgG levels to SARS-CoV-2 S protein at 28 days post-booster vaccination for pediatric participants in the Immunogenicity Population overall and by age cohort, regardless of serostatus at baseline and pre-booster vaccination, compared with that observed at 28 days post-booster vaccination in young adult participants 18 to < 26 years of age.
Serum IgG levels to SARS-CoV-2 S protein, post booster, by age cohort, regardless of serostatus at baseline and pre-booster | Day 0 to Day 28
  Serum IgG levels to SARS-CoV-2 S protein at 28 days post-booster for pediatric participants in the Immunogenicity Population overall and by age cohort, regardless of serostatus at baseline and pre-booster, compared with that observed in pediatric participants at baseline (Day 0).
Serum IgG levels to SARS-CoV-2 S protein , post booster, by age cohort, regardless of serostatus at baseline and pre-booster | Day 0 to Day 35
  Serum IgG levels to SARS-CoV-2 S protein at 28 days post-booster for pediatric participants in the Immunogenicity Population overall and by age cohort, regardless of serostatus at baseline and pre-booster, compared with that observed in pediatric participants at Day 35,
Neutralizing antibody response for pediatric participants and adult participants expressed as Geometric Mean Titers (GMT) | Day 35
  Neutralizing antibody response for pediatric participants compared with adult participants 18 to < 26 years of age from the Adult Main Study at Day 35
Neutralizing antibody response for pediatric participants and adult participants expressed as Sero response (SRR) | Day 35
  Neutralizing antibody response for pediatric participants compared with adult participants 18 to < 26 years of age from the Adult Main Study at Day 35
Serum IgG levels to SARS-CoV-2 S protein after second injection of the initial vaccination series | Day 35
  Serum IgG levels to SARS-CoV-2 S protein 14 days after second injection of the initial vaccination series (Day 35) in pediatric participants in the Immunogenicity Population by age cohort and subsets with and without anti-NP antibodies at baseline.
Treatment and severity of COVID 19 after a PCR-confirmed case | Day 0 to Day 730
  Description of course, treatment and severity of COVID 19 reported after a PCR-confirmed case via the Case Form.
Antibodies to SARS-CoV-2 NP, regardless of whether the infection was symptomatic. | Day 0 to Day 730
  Antibodies to SARS-CoV-2 NP, regardless of whether the infection was symptomatic. Antibodies to SARS-CoV-2 NP at Days 0 and 35, at Crossover Visit 1, at Booster vaccination visit, and at Months 12 and 24 will be used to determine natural infection and to determine the incidence of asymptomatic infection acquired during study follow-up.
Serum IgG levels to SARS-CoV-2 S protein expressed as GMT | Day 180 to Day 730
  Serum IgG levels to SARS-CoV-2 S protein at Months 6 (pre- booster), 7/8 (1-month post-booster), 12, and 24 post-vaccination with NVXCoV2373.
MN titers to SARS-CoV-2 S protein expressed as GMT | Day 180 to Day 730
  MN titers at Months 6 (pre- booster), 7/8 (1-month post-booster), 12, and 24 post-vaccination with NVXCoV2373.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (94):
- United States (47):
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - Coast Clinical Research, LLC, Bellflower, California
  - Apex Research Group, Fair Oaks, California
  - Ark Clinical Research, Long Beach, California
  - Orange County Research Institute, Ontario, California
  - California Research Foundation, San Diego, California
  - Clinical Research of California, Walnut Creek, California
  - Imagine Research of Palm Beach County, Boynton Beach, Florida
  - Palm Harbor Dermatology PA, Brandon, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Cordova Research Institute, LLC, Miami, Florida
  - ARS-Nona Pediatric Center, Orlando, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Tekton Research - Atlanta, Chamblee, Georgia
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - Michael W. Simon, M.D., PSC, Lexington, Kentucky
  - Bluegrass Clinical Research, Inc./All Children Pediatrics, Louisville, Kentucky
  - Velocity Clinical Research - Covington, LA, Covington, Louisiana
  - Velocity Clinical Research - Covington, Covington, Louisiana
  - Velocity Clinical Research - Lafayette LA, Lafayette, Louisiana
  - Craig A. Spiegel, M.D., Bridgeton, Missouri
  - Boeson Research, Missoula, Montana
  - Meridian Clinical Research, Lincoln, Nebraska
  - Be Well Clinical Studies, LLC, Lincoln, Nebraska
  - Corning Center for Clinical Research, Horseheads, New York
  - Velocity Clinical Research, Beachwood, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Lynn Institute of Tulsa, Tulsa, Oklahoma
  - Velocity Clinical Research Grants Pass, Grants Pass, Oregon
  - Tribe Clinical Research, Greenville, South Carolina
  - WR - ClinSearch, LLC, Chattanooga, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Tekton Research Beaumont, Beaumont, Texas
  - PanAmerican Clinical Research, Brownsville, Texas
  - South Texas Clinical Research, Corpus Christi, Texas
  - Bay Colony Pediatrics, Dickinson, Texas
  - Trio Clinical Trials, Houston, Texas
  - Mercury Clinical Research, Houston, Texas
  - Research Your Health, Plano, Texas
  - Mercury Clinical Research - Pediatric Center, Richmond, Texas
  - Tekton Research, San Antonio, Texas
  - Alliance for Multispecialty Research, Layton, Utah
  - Alliance for Multispecialty Research c/o Wee Care Pediatrics - Roy, Roy, Utah
  - Velocity Clinical Research - West Jordan, West Jordan, Utah
  - Clinical Research Partners, LLC, Richmond, Virginia
- Colombia (6):
  - Fundacion Centro de Investigacion Clinica - CIC, Medellín, Antioquia
  - Clinica de la costa, Barranquilla, Atlántico
  - Centro de Atencion e Investigacion Medica S.A.S-CAIMED, Puente Aranda, Bogota D.C.
  - Centro de Atencion e Investigacion Medica - CAIMED, Yopal, Casanare Department
  - Fundacion Oftalmologica de Santander - FOSCAL, Floridablanca, Santander Department
  - Centro de Estudios en Infectologia Pediatrica S.A.S.CEIP, Cali, Valle del Cauca Department
- Dominican Republic (5):
  - PROBEBE en Hospital Universitario Maternidad Nuestra Senora de la Altagracia, Santo Domingo, Nacional
  - Instituto Dermatologico y Cirugia de Piel Dr. Huberto Bogaert Diaz IDCP, Santo Domingo, Nacional
  - MEDYVAC INTERNACIONAL SRL en Clinica Cruz Jiminian, Santo Domingo, Nacional
  - Registrum Group (Hospital Regional Marcelino Velez), Santo Domingo, Nacional
  - Registrum Group (Hospital Materno Infantil San Lorenzo de Los Mina), Santo Domingo, Nacional
- Guatemala (3):
  - Centro de Investigaciones Pediátricas (CIP), Guatemala City
  - SMI (Servicios Medicos Integrales), Guatemala City
  - CECLISA, Guatemala City
- Honduras (3):
  - DEMEDICA, San Pedro Sula, Cortés Department
  - Inverime S.A., Tegucigalpa, Francisco Morazán Department
  - Investigacion Sin Limites, Tegucigalpa, Francisco Morazán Department
- Mexico (8):
  - Panamerican Clinical Research S.A de C.V., Guadalajara, Jalisco
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Tlalpan, Mexico City
  - Innovacion y Desarrollo en Ciencias de la Salud (IDeCSa), Tlalpan, Mexico City
  - Panamerican Clinical Research, Mexico S.A de C.V., Cuernavaca, Morelos
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatan S.C.P., Mérida, Yucatán
  - Panamerican Clinical Research Mexico S.A. de C.V. (Queretaro Site), Querétaro
  - Clinical Research Institute S.C., Tlalnepantla
  - FAICIC S. de R.L. de C.V., Veracruz
- Philippines (6):
  - University of the Philippines Manila - National Institutes of Health (NIH) - Institute of, San Juan City, Batangas
  - Manila Doctors Hospital, Manila, National Capital Region
  - University of the Philippines - Philippine General Hospital, Manila, National Capital Region
  - National Children's Hospital, Quezon City, National Capital Region
  - FEU-NRMF, Quezon City, National Capital Region
  - Medical Mission Group Hospital-Lucban and Southern Luzon State University, Lucena City, Quezon
- South Africa (10):
  - REIMED Riger Park, Boksburg, Gauteng
  - Setshaba Research Centre, Ga-Tshwene, Gauteng
  - Soweto Clinical Trials Centre, Johannesburg, Gauteng
  - WiWits RHI - Shandukani Research Centre, Johannesburg, Gauteng
  - Wits Vida Nkanyezi Site- Rahima Moosa Mother and Child Hospital, Johannesburg, Gauteng
  - Wits Vida- Chris Hani Baragwanath Hospital, Soweto, Gauteng
  - Limpopo Clinical Research Initiative, Thabazimbi, Limpopo
  - Tiervlei Trial Centre, Bellville, Western Cape
  - Be Part Yoluntu Centre - Paarl, Paarl, Western Cape
  - Stellenbosch University Worcester, Worcester, Western Cape
- Spain (4):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (2):
  - Lakeside Healthcare Research, Corby, Northamptonshire
  - St Georges Hospital, London